CLINICAL TRIAL: NCT02167659
Title: A Randomized Trial Evaluating Bioimpedance Spectroscopy Versus Tape Measurement in the Prevention of Lymphedema Following Locoregional Treatment for Breast Cancer (PREVENT)
Brief Title: Bioimpedance Spectroscopy Versus Tape Measure in Prevention of Lymphedema (PREVENT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ImpediMed Limited (Industry)
Collaborators: Vanderbilt University (Other); Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VICCBRE1438
Record Dates: First submitted 2014-06-12; First posted 2014-06-19 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Lymphedema
Keywords: Lymphedema; Breast cancer; Bioimpedance Spectroscopy; L-Dex
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIS Assessment (Experimental): Patients will undergo measurements by trained staff. Measurements will be performed pre-op and at 3, 6, 12, 15*, 18, 21*, 24, and 36 months post-op. Measures include L-Dex, skin assessment and self-report forms. Patients with < 6.5 L-Dex units change will continue follow-up for 36 months. Patients with an L-Dex value change ≥ 6.5 will undergo circumference measurement and begin treatment for 4 weeks with a 23-32 mmHg compression sleeve with gauntlet. At the end of 4 weeks patients will have their arms measured. Those demonstrating improvement will continue with follow up. Those not demonstrating improvement will be removed from the study and their medical oncologist or surgeon will be notified.
  *At discretion of the site PI or attending physicians.
  Interventions: Device: 23-32 mmHg compression sleeve with gauntlet
- Tape Measure (Active Comparator): Patients will undergo measurements by trained staff. Measurements will be performed pre-op and at 3, 6, 12, 15*, 18, 21*, 24, and 36 months post-op. Measures include arm volume (tape measure), skin assessment and self-report forms. Patients with no volume increase will continue follow-up for 36 months. Patients with a volume change of between ≥ 5% and < 10% in the at-risk limb will undergo L-Dex testing and begin treatment for 4 weeks with a 23-32 mmHg compression sleeve with gauntlet. At the end of 4 weeks patients will have their arms measured. Those demonstrating improvement will continue with follow up. Those not demonstrating improvement will be removed from the study and their medical oncologist or surgeon will be notified.
  *At discretion of the site PI or attending physicians.
  Interventions: Device: 23-32 mmHg compression sleeve with gauntlet

INTERVENTIONS:
Device: 23-32 mmHg compression sleeve with gauntlet — A compression intervention consisting of a sleeve and gauntlet with 23-32mm of tension worn for four weeks that is initiated based on a BIS L-Dex change that is ≥6.5 units higher than pre-surgical baseline measure, or a tape measurement guided volume change in the affected arm that is between ≥5% and <10% above pre-surgical baseline.
  Other Names: mediven harmony

SUMMARY:
Based upon the current state of science, the investigators are proposing to conduct a randomized clinical trial in which participants are randomized post-surgery to either BIS or circumferential (tape) measurements for follow-up arm measurements. When patients in the BIS group have an L-Dex change that is ≥6.5 units higher than the pre-surgical baseline measure, and when patients in the tape measurement group have a volume change in the at-risk arm that is between ≥ 5% and <10% above pre-surgical baselines (without similar change in non-at-risk arm), both will receive four weeks of 23-32 mm compression sleeve and gauntlet therapy.

DETAILED DESCRIPTION:
The treatment of lymphedema following breast cancer therapy is typically a burdensome multi-modality process that entails different degrees of intensity depending on the severity of fluid accumulation. In breast cancer survivors, it is most commonly initiated after visible swelling occurs in a limb. Common treatments utilized are multi-modality and include massage, compression, exercises, and skin care. The current gold standard treatment for advanced fluid accumulation is complex decongestive physiotherapy (CDP). CDP includes components of compression, lymphatic drainage, skin care, and exercise and is commonly delivered in two phases with the first phase being a several week course delivered in the outpatient clinical setting and the second a home maintenance program. CDP is considered the gold standard due to prospective data demonstrating its efficacy, a series of 537 patients found significant arm volume decreases with CDP and subsequent studies have confirmed volume reductions along with improved quality of life in those patients undergoing CDP. Studies comparing CDP to other treatment modalities are limited but some have favored CDP. CDP is limited in that access to long term prospective follow-up treatment may not take place and it requires significant resources and costs.

Recent studies have suggested that early diagnosis and treatment allow for less burdensome and aggressive therapy utilization moving forward. Increasing data support the idea that early intervention improves outcomes for women with lymphedema following breast cancer treatment. Recent prospective data have shown that with a short course of compression therapy (sleeve and gauntlet), ranging from 4 to 6 weeks, the rate of progression of fluid accumulation is limited. Specifically, the Stout Gergich et al. study provided sound preliminary data to support that four weeks of treatment using a 20-30 mmHg compression garment and gauntlet can, over 18 months of post intervention follow-up, reduce volume and prevent the need for CDP.

These findings are encouraging; however, it should be noted that these studies have significant limitations including small patient numbers, limited follow up, a lack of randomization, and a lack of subclinical detection of increasing extracellular fluid. Therefore, while some data exist that suggest that early intervention with clinically apparent extracellular fluid accumulation is beneficial, there are less data to support the hypothesis that subclinical detection and subsequent early intervention are beneficial. Based on data from these studies, it may be possible to prevent chronic lymphedema with early detection and intervention. Early detection may be best achieved by identifying changes in extracellular fluid instead of change in whole arm volume. Given the potential to improve patient outcomes and possibly prevent chronic lymphedema, additional research is warranted in large randomized trials that address some of the limitations of the previous work.

BIS is a technology designed to identify changes in extracellular fluid. The investigators propose to determine if subclinical detection of increasing extracellular fluid via BIS and subsequent early treatment with four weeks of a compression sleeve and gauntlet results in a reduction in the rates of progression to chronic lymphedema as compared to the same intervention when initiated from use of the most common arm measurement method (tape measurement).

The investigators will secondarily explore selective correlatives related to lymphedema and lymphedema progression. As multiple factors may lead to lymphedema, the influence of potential risk factors on lymphedema progression will be evaluated. Time to actual progression will also be examined. Because lymphedema results in problematic symptoms and diminished quality of life, correlatives using validated instruments will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer or Ductal Carcinoma In Situ (DCIS)
* Planned surgical procedure
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior history of breast cancer, breast/chest wall/axillary radiation therapy
* Definitive breast surgical procedure prior to enrollment.
* Active implanted medical device (e.g., cardiac pacemakers, defibrillators) or patients connected to electronic life support devices or metallic devices that would interfere with BIS measurements.
* Conditions that could cause swelling (e.g., pregnancy, congestive heart failure, chronic/acute renal disease, cor pulmonale, nephrotic syndrome, nephrosis, liver failure or cirrhosis, pulmonary edema, and thrombophlebitis, or deep vein thrombosis in arms
* Previous treatment for lymphedema of either arm.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, or cardiac arrhythmia.
* Psychiatric illness (e.g., diagnosed schizophrenia or documented dementia) that would limit compliance with study requirements.
* Known allergy to electrode adhesives or woven knit compression fabrics
* Bilateral breast cancer or planned bilateral mastectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1201 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of progression of lymphedema | 3 years
  To determine if subclinical detection of extracellular fluid accumulation via bioimpedance spectroscopy and subsequent early intervention reduce the rate of progression to CDP relative to rates seen using standard tape measurements.

SECONDARY OUTCOMES:
Number of participants with risk factors associated with lymphedema. | 3 years
  To evaluate factors associated with progression requiring CDP (e.g., Body Mass Index (BMI), Seroma, Smoking, Age, Air Travel).
Time elapsed between identification of increasing fluid and referral out of study for continued swelling. | 3 years
  To evaluate time to progression requiring CDP.
Number of participants with improved skin condition, symptoms and quality of life. | 3 years
  To determine if subclinical detection of extracellular fluid accumulation and subsequent early intervention improves skin condition, symptoms, and quality of life compared with standard tape measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila H Ridner, PhD, Principal Investigator — Vanderbilt University
Locations (10):
- United States (9):
  - Mayo Clinic, Jacksonville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Southeast Health, Cape Girardeau, Missouri
  - New York Presbyterian - University Hospital of Columbia and Cornell, New York, New York
  - Allegheny Health Research Institute, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Massey Cancer Center, Richmond, Virginia
- Macquarie University, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boyages J, Vicini FA, Manavi BA, Gaw RL, Koelmeyer LA, Ridner SH, Shah C. Axillary Treatment and Chronic Breast Cancer-Related Lymphedema: Implications for Prospective Surveillance and Intervention From a Randomized Controlled Trial. JCO Oncol Pract. 2023 Dec;19(12):1116-1124. doi: 10.1200/OP.23.00060. Epub 2023 Oct 10. PMID 37816208
- [Derived] Dietrich MS, Gaitatzis K, Koelmeyer L, Boyages J, Abramson VG, McLaughlin SA, Ngui N, Elder E, French J, Hsu J, Hughes TM, Stolldorf DP, Shah C, Ridner SH. Prospective Surveillance with Compression for Subclinical Lymphedema: Symptoms, Skin, and Quality-of-Life Outcomes. Lymphat Res Biol. 2023 Jun;21(3):304-313. doi: 10.1089/lrb.2022.0020. Epub 2022 Sep 20. PMID 36126315
- [Derived] Ridner SH, Dietrich MS, Boyages J, Koelmeyer L, Elder E, Hughes TM, French J, Ngui N, Hsu J, Abramson VG, Moore A, Shah C. A Comparison of Bioimpedance Spectroscopy or Tape Measure Triggered Compression Intervention in Chronic Breast Cancer Lymphedema Prevention. Lymphat Res Biol. 2022 Dec;20(6):618-628. doi: 10.1089/lrb.2021.0084. Epub 2022 Jan 28. PMID 35099283